CLINICAL TRIAL: NCT06976944
Title: Randomized Phase II Study of Pembrolizumab + Paclitaxel +/- Bevacizumab in Patients With Recurrent Triple-Negative Breast Cancer Who Received Perioperative Immunotherapy
Brief Title: Pembrolizumab + Paclitaxel +/- Bevacizumab for Triple-negative Breast Cancer
Acronym: PRELUDE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yukinori Ozaki (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Yukinori Ozaki, Director of Breast Medical Oncology, Japanese Foundation for Cancer Research
Organization: Japanese Foundation for Cancer Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJOG16522B; jRCT2031250076 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Triple-Negative Breast Cancer
Keywords: Recurrent Triple-Negative; Breast Cancer; checkpoint inhibitor; angiogenesis inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab + paclitaxel + bevacizumab (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Bevacizumab
- Pembrolizumab + paclitaxel (Active Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Protocol treatment will continue until worsening of the participant's underlying disease or unacceptable toxicity is observed or the participant withdraws the consent, or the participant meets other discontinuation criteria.
  Pembrolizumab: Intravenous infusion(400 mg/body, every 6 weeks starting on Day 1 of Cycle 1)
Drug: Paclitaxel — Protocol treatment will continue until worsening of the participant's underlying disease or unacceptable toxicity is observed or the participant withdraws the consent, or the participant meets other discontinuation criteria.
  Paclitaxel: Intravenous infusion(90 mg/m^2, on Days 1, 8, and 15, starting on Day 1 of Cycle 1 with a 28-day cycle)
Drug: Bevacizumab — Protocol treatment will continue until worsening of the participant's underlying disease or unacceptable toxicity is observed or the participant withdraws the consent, or the participant meets other discontinuation criteria.
  Bevacizumabl: Intravenous infusion(10 mg/kg, on Days 1, and 15, starting on Day 1 of Cycle 1 with a 28-day cycle)
  Arms: Pembrolizumab + paclitaxel + bevacizumab

SUMMARY:
* Breast cancer is histologically divided into non-invasive (approximately 10%) and invasive (approximately 90%), with invasive cancer being the target of chemotherapy. Invasive carcinoma is classified into four subtypes according to the expression levels of hormone receptor (HR) and human epidermal growth factor receptor type 2 (HER2). Among them, triple negative breast cancer accounts for 10% of invasive cancers and is the subtype with the poorest prognosis.
* For triple negative breast cancer that is operable, chemotherapy with pembrolizumab is administered either preoperatively or postoperatively (perioperative period). For recurrent triple negative breast cancer , combination chemotherapy with multiple agents is the standard of care, especially in the case of PD-L1-positive patients, chemotherapy with an immune checkpoint inhibitor related to PD-1 (pembrolizumab or atezolizumab) is administered.
* Although the KEYNOTE355 trial demonstrated the efficacy of pembrolizumab plus paclitaxel therapy in patients with PD-L1-positive triple negative breast cancer in postoperative relapse, this trial did not include patients who received pembrolizumab in the perioperative period. Therefore, it is not known if there is any benefit to re-administering pembrolizumab to these patients after relapse.
* Bevacizumab is used as standard therapy for triple negative breast cancer in combination with paclitaxel. Bevacizumab itself is an anti-tumor agent that inhibits angiogenesis, but has also been reported to activate immunity against cancer, suggesting that it may enhance the effect of pembrolizumab.

Based on the above, the investigators planned this trial to evaluate whether pembrolizumab + paclitaxel + bevacizumab therapy is more effective than pembrolizumab + paclitaxel therapy in PD-L1-positive triple negative breast cancer patients who relapse after receiving immune checkpoint inhibitors in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are 18 years of age or older on the day of signing informed consent with histologically or cytologically confirmed diagnosis of invasive breast cancer will be enrolled in this study.
2. Participants have been confirmed to be ER negative, HER2 negative according to the latest ASCO/CAP criteria. However, it does not matter whether the result is positive or negative for PgR.
3. Participants have been confirmed to be PD-L1 positive in each site's evaluation using biopsy specimen or surgical specimen.
4. Participants who have not undergone chemotherapy for recurrent breast cancer. However, prior treatment of Olaparib for metastatic recurrence or unresectable advanced cancer in participants with BRCA gene pathogenic variant is allowed.
5. Participants must have recurred after treatment with an anti-PD-1/PD-L1 antibody administered as monotherapy or in combination with other ICIs or chemotherapies as a perioperative drug therapy for triple negative breast cancer.
6. Have an Eastern Cooperative Oncology Group performance status of 0 to 1.

Exclusion Criteria:

1. Participants with progressive disease on RECIST or clinically diagnosed during preoperative ICI and chemotherapy.
2. Known additional malignancy that is progressing or has required active treatment within the past 3 years prior to enrollment.
3. Has known active CNS metastases and/or carcinomatous meningitis.
4. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Through protocol treatment discontinuation, approximately 9 months

SECONDARY OUTCOMES:
Overall response rate | Through protocol treatment discontinuation, approximately 9 months
Overall survival | Through study completion, approximately 3.5 years
Disease control rate | Through protocol treatment discontinuation, approximately 9 months
Incidence of adverse events | Until 1 month after protocol treatment discontinuation, approximately 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Toshimi Takano, Study Chair — Cancer Institute Hospital of JFCR
Locations (15):
- Japan (15):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Gifu University Hospital, Gifu, Gifu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Kindai University Hospital, Sayama-shi, Osaka
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - SHOWA Medical University Hospital, Shinagawa-ku, Tokyo